CLINICAL TRIAL: NCT01369030
Title: Deplin® P.L.U.S. Program (Progress Through Learning Understanding & Support)
Status: Completed | Type: Observational
Sponsor: Pamlab, Inc. (Industry)
Collaborators: InfoMedics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D-009
Record Dates: First submitted 2011-05-17; First posted 2011-06-08 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Major Depressive Disorder
Keywords: L-methylfolate; Deplin; depression; antidepressant; combination therapy; augmentation; folate; folic acid; homocysteine; methionine; MTHFR genotype; C677T mutation; vitamin B6; vitamin B12
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — 5-methyltetrahydrofolate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Deplin®: Subjects with depression who have been prescribed Deplin® daily.
  Interventions: Other: Deplin®

INTERVENTIONS:
Other: Deplin® — Deplin® is an orally administered medical food available in a 7.5mg tablet or a 15mg caplet with each containing either 7.5mg or 15mg of L-methylfolate, respectively - which is the primary biologically active and immediately bioavailable form of folate. Dosage for this study will be 1 15mg caplet QD.

SUMMARY:
This study will be an observational study in which patients who have been prescribed Deplin® are invited to participate in surveys regarding their experiences with Deplin®. The purpose of this study is to increase the understanding of the role of L-methylfolate among patients who are candidates for Deplin®, provide patients with personalized education and support, and contribute to the overall understanding of the needs and concerns of patients being treated for depression.

DETAILED DESCRIPTION:
Surveys used to conduct this study will be administered via telephone or online by InfoMedics, Inc., a company with a system for developing such patient-physician feedback programs. Participating physicians will ask their patients to participate in the program after Deplin® has been prescribed and provide them with a brochure containing an introduction to the program and instructions on how to enroll. Patients self-enroll, take a brief survey before starting their Deplin® prescription, and then a follow-up survey after 90 days of treatment with Deplin®. As patients complete surveys within the study, their physician will receive individualized feedback reports outlining their patient's treatment experience and progress. Patients will also receive a copy of their own reports, to help encourage them to continue taking Deplin® as directed. Patients will also receive educational materials about managing their depression.

ELIGIBILITY:
Inclusion Criteria:

* New Deplin® Start
* Only for patients with depression who have been prescribed brand name Deplin® to help metabolic management of depression.
* Clinically depressed patients who have been prescribed Deplin® in combination with an antidepressant.
* At the start of antidepressant therapy
* As augmentation to antidepressant therapy

Exclusion Criteria:

* Patients who do not meet DSM IV criteria for major depression
* If participant indicates that he or she did not get a prescription for Deplin®, he/she will not be able to complete the survey(s).
* For follow-up surveys, if the participant indicates that he/she has not been taking Deplin®, he/she will not be able to complete the survey(s).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Depression Who Have Been Prescribed Deplin®
Sampling Method: Probability Sample
Enrollment: 554 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Shelton, M.D., Principal Investigator — Vanderbilt University School of Medicine; Sloan Manning, M.D., Principal Investigator — Mood Disorders Clinic at Moses Cone Family Practice Center
Locations (2):
- United States (2):
  - Moses Cone Family Practice Center, Greensboro, North Carolina
  - Vanderbilt University School of Medicine, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2010 and January 2012, patients of at least 18 years of age who had been prescribed Deplin® by their physician for the treatment of major depression were offered to participate in the study by their prescibing physician, consisting of about 550 participating physicians located at various clinical sites country-wide.
Pre-assignment Details: Participants may have excluded themselves from the overall study after self-enrolling in the program if they did not complete the designated surveys prior to using Deplin® (Baseline) or at the 90-day time point post-treatment initiation.
Period: Overall Study
Arm/Group | Deplin®
Started | 594
Completed | 554
Not Completed | 40

BASELINE CHARACTERISTICS:
Population: A total of 594 completed the baseline and follow-up surveys and of those only 554 with a baseline PHQ-9>=5 were included in the analysis. Majority of the participants were female, and the study was approximately equal distribution across the four depression severity groups of interest.
Arm/Group | Deplin®
Number analyzed (Participants) | 554
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 470
  >=65 years | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (14.1)
Gender [Number; unit: participants] — Baseline gender characteristic categories include female, male, and unknown. 16 enrolled subjects were listed as unknown.
  participants
    Female | 424
    Male | 114
Region of Enrollment [Number; unit: participants]
  United States | 554

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression Severity as Measured by the 9-item Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 is a depression scale used to assess brief depression severity by rating symptoms and functional impairment experienced in the last two weeks. The questionnaire contains a total of 9 questions, and each question is scored on a range from 0-3. The minimum value "0" represents not at all, "1" several days, "2" indicates more than half the days, and the maximum value "3" stands for nearly every day. The total possible range is 0-27. The total number of each 0, 1, 2, 3 is added and multiplied by its value (0=0, 1=1, etc.) to produce a total score generated from the subtotal sum. The PHQ-9 total score is interpreted as follows: 0-4 represents minimal depression, 5-9 as mild depression, 10-14 as moderate depression, 15-19 moderately severe depression, and 20-27 severe depression.
Time Frame: Baseline to Endpoint (90 days)
Population: Analyses were performed on the 554 patients who had a baseline PHQ-9>=5 and further analyzed by baseline depression severity groups defined by baseline PHQ-9 scores: 5<=PHQ-9<=9; 10<=PHQ-9<=14; 15<=PHQ-9<=19; and 20<=PHQ-9<=27.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deplin®
Number analyzed (Participants) | 554
units on a scale
  Mean baseline PHQ-9 Score | 14.6 (5.8)
  Mean endpoint PHQ-9 Score | 6.1 (5.0)
  Mean reduction in PHQ-9 Score | 8.5 (6.3)
Statistical Analysis 1: Comparison: Deplin®; Test type: Superiority or Other; p = 0.000, Wilcoxon signed-rank test; Mean Difference (Net) = 8.5, Standard Deviation 6.3

2. Secondary Outcome: Proportion of Patients Reporting Difficulty in Daily Functioning Due to Depressive Symptoms
Time Frame: Baseline to Endpoint (90 days)
Measure: Number; unit: percentage of participants
Arm/Group | Deplin®
Number analyzed (Participants) | 554
percentage of participants | 37.5

3. Secondary Outcome: Change in Overall Patient Satisfaction With Deplin® Using a 9-point Satisfaction Scale
Description: Mean satisfaction with medication was rated on 1 to 9 point scale, 1 indicating "not at all satisfied" and 9 as "very satisfied."
Time Frame: Baseline to Endpoint (90 days)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Deplin®
Number analyzed (Participants) | 554
units on a scale | 7.0 [1 to 9]

ADVERSE EVENTS:
Arm/Group | Deplin®
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Patients self-enrolled in the program and data presented was based on self-reported close-ended questions; selection bias may be present for those who chose not to enroll or complete the surveys. No clinical evaluations were conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No